CLINICAL TRIAL: NCT04818580
Title: A Prospective Cohort Study Comparing the Effect of Progressive Tension Sutures and Drains to Drains Alone on Rates of Hematoma and Seroma in Gender Affirming Mastectomy for Transgender Men
Brief Title: Progressive Tension Sutures in Gender Affirming Mastectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of key personnel, difficulties with recruiting.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-01803
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Hematoma; Seroma
Keywords: Mastectomy
MeSH Terms: conditions — Hematoma; Seroma

STUDY DESIGN:
Who Masked: Participant
Masking Description: A random number generator will be used. Subjects will be blinded as to which side of the chest has the sutures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right-Sided Progressive Tension Sutures (Experimental)
  Interventions: Procedure: Progressive Tension Sutures
- Left-Sided Progressive Tension Sutures (Active Comparator)
  Interventions: Procedure: Progressive Tension Sutures

INTERVENTIONS:
Procedure: Progressive Tension Sutures — In each patient, one side of the chest will receive progressive tension sutures inside the mastectomy pocket, from pectoral fascia to underside of mastectomy flap. 2-0 Vicryl about 15-20 sutures per chest. Both sides will receive bilateral drains (standard of care)

SUMMARY:
50 patients seeking gender affirming mastectomy will be treated with different closure techniques in each side of their chest - one side will receive progressive tension sutures between pectoral fascia and the mastectomy flap, and the other side will not. Both sides will have drains in the mastectomy site. Rates of hematoma, seroma, and other complications will be compared between each chest side via standard statistical techniques for hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

1. Being consulted for gender affirming mastectomy with the senior author (AH).
2. >18 years of age at the time of enrollment.
3. Transgender or gender nonbinary gender identity.
4. All co-morbidities and all indications.

Exclusion Criteria:

1. Age less than 18 years.
2. BMI < 23.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender men
Enrollment: 3 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Total volume of Drain Fluid | Visit 2, Day 7
  Participants will record drain outputs each time they empty drains in the Postoperative Drain Output Record (mL)
Total volume of Drain Fluid | Visit 3, Day 14
  Participants will record drain outputs each time they empty drains in the Postoperative Drain Output Record (mL)
Total volume of Drain Fluid | Visit 4, Day 30
  Participants will record drain outputs each time they empty drains in the Postoperative Drain Output Record (mL)

CONTACTS AND LOCATIONS:
Overall Officials: Alexes Hazen, MD FACS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Thomas.Calahan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.